CLINICAL TRIAL: NCT06917521
Title: EARLY IDENTIFICATION OF VENTILATOR ASSOCIATED PNEUMONIA USING MACHINE LEARNING TECHNIQUES: A PROSPECTIVE COHORT
Brief Title: VAP Identification by AI
Acronym: AI-VAP
Status: Completed | Type: Observational
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-00624 CE 4085
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Ventilator Associated Pneumonia ( VAP)
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ventilator-associated pneumonia (VAP) is the most frequent infection in the intensive care setting. For VAP there is currently no reliable diagnostic criteria. We aimed with the present study, using data from the mechanical ventilator to identify early this infection using artificial intelligence methods .

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is defined as a hospital-acquired pneumonia occurring in patients submitted to invasive mechanical ventilation (MV) for at least 48 hours. VAP represents the most prevalent nosocomial infection in the intensive care setting. VAP is burdened by prolonged duration of MV and hospital length of stay and consequently increases hospital costs. Moreover, mortality and antibiotic use are also significantly affected. Unfortunately, there is currently no valid, accurate diagnostic criteria of VAP because even the most widely used ones are neither sensitive nor specific.. The insufficient sensitivity of these criteria to rule out VAP carries the risk of antibiotic overuse with the consequently emerging of antibiotic resistance and superinfections. On the other hand, the insufficient specificity to rule in VAP carries the risk of delayed administration of antimicrobial therapy leading to increased mortality. Ventilator-associated event surveillance failed to accurately identify VAP, too . The purpose of the present study is to develop different AI-algorithms using data continuously recorded form the mechanical ventilator in supporting clinicians for the early detection of VAP. An accurate AI-algorithm for early VAP identification has the potential to reduce morbidity, mortality, exposure to broad-spectrum and/or unnecessary antibiotics and finally to reduce costs.

ELIGIBILITY:
Inclusion Criteria:

* adult patients admitted to our ICU requiring invasive respiratory support for at least 48 hours

Exclusion Criteria:

* previuos pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients admitted to our ICU requiring invasive respiratory support for at least 48 hours will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Early identification of VAP | From July 2023 to Mars 2025
  Sensitivity, specificity, AUROC and AUPRC

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale civico Lugano, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided